CLINICAL TRIAL: NCT07044388
Title: Coping With Asthma Throughout Life Management: CALM Program for African American Adult Patients With Asthma
Brief Title: Coping With Asthma Throughout Life Management Program
Acronym: CALM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: Pro00114349
Record Dates: First submitted 2025-06-23; First posted 2025-07-01 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-06

CONDITIONS: Asthma; Stress
MeSH Terms: conditions — Asthma | interventions — Coping Skills

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Randomized (Experimental): Group will receive intervention method
  Interventions: Behavioral: Coping with asthma through life management program
- Waitlist Control Group (Other): Participants will receive no intervention (control) during the trial. However, after the study is completed, they will have the option to receive intervention.
  Interventions: Behavioral: Waitlist Control (CALM)

INTERVENTIONS:
Behavioral: Coping with asthma through life management program — Participants will complete surveys, learn stress coping strategies, receive asthma education information, and obtain access local community financial resources.
  Arms: Randomized
Behavioral: Waitlist Control (CALM) — Participants in this group will complete surveys but will not receive the CALM intervention. Upon completing the study after 12 weeks they will be able to complete the program if they would like the resources/materials to learn healthy stress coping strategies, asthma health education, and access to financial resources.
  Arms: Waitlist Control Group

SUMMARY:
The purpose of this study is to determine if the Coping with Asthma through Life Management (CALM) intervention, designed to help Black adult with asthma cope with stress, is feasible and acceptable.

DETAILED DESCRIPTION:
Asthma medication nonadherence is a major contributor to asthma morbidity and mortality in Black adults. Black adults with asthma reported that increased psychosocial stress (e.g., perceived discrimination, job stress, caregiver burden), health-related stress (e.g., concern about asthma control), and economic stress (e.g., economic strain) were barriers to asthma medication adherence and control. The study's hypothesis is that CALM, targeting multiple stressors specifically faced by Black adults with asthma, will be feasibly implemented in a health system, will be acceptable to program participants, and will be a potentially effective intervention to improve asthma medication adherence and asthma control.

ELIGIBILITY:
Inclusion Criteria:

* At least the age of 18
* Self identify as Black/African-American
* Self-report current asthma diagnosis
* Asthma must be persistent (Prescribed an inhaled corticosteroid (alone or in combination)
* Asthma must be uncontrolled (≥1 exacerbation in the past years OR Asthma Control Questionnaire > 0.75)
* Have moderate-high stress (Perceived Stress Scale ≥ 14)
* Presented at any Primary Care clinic in the past 3 years.

Exclusion Criteria:

* Unable or unwilling to give consent
* Diagnosis of a psychotic disorder
* Positive responses to questions regarding suicidality

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-12-18 (Estimated); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Intervention Measure (FIM) | 12 weeks
  The FIM has four items and the total score ranges from 4 to 20, where a higher score indicates greater feasibility.
Acceptability of Intervention Measure (AIM) | 12 Weeks
  The AIM has four items and the total score ranges from 4 to 20, where a higher score indicates greater acceptability.
Intervention Appropriateness Measure (IAM) | 12 Weeks
  The IAM has four items and the total score ranges from 4 to 20, where a higher score indicates greater appropriateness.

SECONDARY OUTCOMES:
Asthma Control Questionnaire (ACQ-6) | 1 week
  The ACQ-6 is a six-question questionnaire used to assess asthma control, focusing on symptoms and rescue medication use. Scores range from 0 to 6, with lower scores indicating better asthma control. A score of 1.5 or higher suggests poorly controlled asthma.
Perceived Stress Scale (PSS-10) | 1 month
  The PSS-10 is a 10-item questionnaire that evaluates the degree to which an individual has perceived life as unpredictable, uncontrollable, and overloading over the previous month. Scores range from 0 to 40, with higher scores indicating higher levels of perceived stress.
Asthma Quality of Life Questionnaire, Marks (AQLQ-M) | 2 weeks
  The AQLQ-M is a 20-item self-administered questionnaire to measure quality of life in adults with asthma. Scores range from 20 to 100, with higher scores indicating a greater negative impact of asthma.
Number of participants with an asthma exacerbation event | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Isaretta Riley, MD-MPH, Principal Investigator — Duke University

IPD SHARING:
Plan to Share IPD: No